CLINICAL TRIAL: NCT00843570
Title: A Randomised Controlled Trial of Natural Versus Hormone Replacement Therapy Cycles in Frozen Embryo Replacement IVF: a Pilot Study
Brief Title: Natural Versus HRT Cycles in Frozen Embryo Replacement Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Fertility Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER01; EudraCT 2009-009323-11
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
Keywords: IVF; Frozen Embryo Replacement
MeSH Terms: conditions — Infertility | interventions — Nafarelin; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Natural FER (frozen embryo replacement)
- 2 (Active Comparator): HRT-FER (Down regulated frozen embryo replacement)
  Interventions: Drug: Nafarelin acetate, Oestradiol Valerate, Progesterone

INTERVENTIONS:
Drug: Nafarelin acetate, Oestradiol Valerate, Progesterone — Nafarelin acetate, Nasal spray, 400 mcg b.d., 4 weeks Oestradiol Valerate, tablet, 2mg o.d day 1-5, 2mg b.d. day 6-9, 2mg t.d.s day 10-13 (step-up protocol), 2mg q.d.s (if pregnancy confirmed, 4-10 weeks Progesterone, pessary, 200mg b.d. and t.d.s. (if pregnancy confirmed), 2-10 weeks
  Other Names: Synarel,Progynova,Cyclogest
  Arms: 2

SUMMARY:
Frozen Embryo Replacement (FER)is a fertility treatment by which stored embryos from a fresh IVF treatment cycle are thawed and transferred into the uterus. Frozen embryos can be replaced either in the middle of a natural menstrual cycle (Natural FER) or in a cycle where the woman takes drugs to suppress her own hormones, and then takes Hormone Replacement Therapy (HRT) to prepare her uterus for the transfer of embryos(HRT - FER).

Both are widely used methods of fertility treatment. However, to date no well designed studies have been reported in which the two methods have been compared. This study aims to compare the two treatments in order to establish the best treatment protocol.

The study design is a single centre open randomized controlled trial funded by the Oxford Fertility Unit.

100 women who are considering FER treatment at the Oxford Fertility Unit and are eligible for the study will be recruited.

After giving their written consent they will be randomised to one of 2 groups: Natural FER and HRT FER.

Patients in both groups will be asked to attend one initial visit, which is additional to patients not taking part in the study.

Subsequent visits will depend on the treatment group but will not be additional for study participants. All visits requiring ultrasound will involve recording 3-D measurements, which increases the length of each visit by approximately 10 minutes. A patient satisfaction questionnaire would be completed at the end of the cycle.

A urinary pregnancy test is performed at home 2 weeks following the embryo transfer visit. If this is positive then further visits to the unit are arranged to confirm the clinical pregnancy.

Inclusion in the study would not increase the length of time of either treatment cycle. Follow up would extend to obtaining pregnancy outcome information.

ELIGIBILITY:
Inclusion Criteria:

* Women attending Oxford Fertility Unit planning a frozen embryo replacement cycle.
* Willing and able to give informed consent for participation in the study.
* Age at original fresh IVF cycle < 40 years old.
* At least 3 embryos frozen in storage
* First or second FER cycle
* Regular ovulatory menstrual cycles, confirmed by luteal progesterone levels >16nmol/L and with cycle length < 35 days.

Exclusion Criteria:

* Women with irregular cycles (outlined above), including amenorrhoea or oligomenorrhoea.
* Co-existing medical illness including renal, cardiac and liver disease
* Women for whom the study medication(s) are contraindicated or who have known allergic reactions to study medication(s)
* Women who have already taken part in this trial (i.e. cannot have more than one treatment cycle as a participant in this trial)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The live birth rate in each group | 22 - 40 weeks following embryo transfer

SECONDARY OUTCOMES:
Clinical pregnancy rates (CPR) | 4 weeks after embryo transfer (at 6/40 pregnancy)
Implantation rate (defined as the number gestational sacs visible on ultrasound divided by the number of embryos replaced and expressed in percentage) | 4 weeks following embryo transfer (6/40 pregnancy)
3D endometrial volume and blood flow indices | various from day 1 to embryo transfer
Patient satisfaction with treatment | 4-10 weeks (at embryo transfer)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Child, MA MD MRCOG, Principal Investigator — Nuffield Department of Obstetrics and Gynaecology, University of Oxford
Locations (2):
- United Kingdom (2):
  - Nuffield Department of Obstetrics and Gynaecology, University of Oxford, Oxford, Oxfordshire
  - Oxford Fertility Unit, Oxford, Oxfordshire

REFERENCES:
- [Derived] Mounce G, McVeigh E, Turner K, Child TJ. Randomized, controlled pilot trial of natural versus hormone replacement therapy cycles in frozen embryo replacement in vitro fertilization. Fertil Steril. 2015 Oct;104(4):915-920.e1. doi: 10.1016/j.fertnstert.2015.07.1131. Epub 2015 Aug 5. PMID 26255087